CLINICAL TRIAL: NCT02324218
Title: Incidence of Hepatitis B Diagnosis Among Diabetes Mellitus Patients of 0-80 Years of Age, in the United Kingdom Clinical Practice Research Datalink (CPRD)
Brief Title: This Study Aims to Determine the Incidence, of Hepatitis B Diagnosis Among Diabetes Mellitus Patients of 0-80 Years of Age
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 201335; 14_114 (Other: Independent Scientific Advisory Committee (ISAC) ID)
Record Dates: First submitted 2014-12-11; First posted 2014-12-24 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Hepatitis B
Keywords: Diabetes mellitus; Hepatitis B; Incidence
MeSH Terms: conditions — Hepatitis B; Diabetes Mellitus | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Diabetes mellitus Group: All the subjects with diabetes mellitus diagnosed with hepatitis B, reported in the CPRD database of UK, from the Year 2000 to 2012.
  Interventions: Other: Data collection
- Non-Diabetes mellitus Group: All the subjects with hepatitis B who are diagnosed negative diabetes mellitus, reported in the CPRD database of UK, from the Year 2000 to 2012.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data extraction from CPRD database of UK.

SUMMARY:
This study is being conducted to assess the risk of hepatitis B (HepB) diagnosis among diabetes mellitus (DM) and non-DM patients of 0-80 years of age with in a large population-based cohort in United Kingdom (UK) using data from the CPRD database.

DETAILED DESCRIPTION:
The study is a retrospective, observational, descriptive, cohort study, in DM and non-DM patients of 0-80 years of age. As a first step the eligible baseline population from CPRD will be defined as per the data quality qualifiers, which include subjects aged 0-80 years, "acceptable for research" registered in practices classified as "up to standard" by the CPRD for the time period 2000- 2012. The following cohorts will be defined from the baseline population:

* DM cohort: Patients diagnosed with type 1 or type 2 DM, as confirmed by diagnosis medical codes with or without a DM related drug or monitoring devices prescription.
* Non-DM cohort: Patients with the absence of personal history of DM diagnosis or antidiabetic drug or monitoring devices prescriptions.

From the above defined cohorts, HepB cases will be identified based on clinical diagnosis codes, Hospital Episodes Statistics (HES) or positive diagnostic laboratory tests results.

ELIGIBILITY:
Inclusion Criteria:

* Subjects, 0 to 80 years of age during the study period.
* Subjects acceptable for research as per CPRD definition:

  * Acceptable flag for research.
* Subjects with at least 12 months of observation time at the time of inclusion in the study:

  * Subjects have to be registered in the CPRD database for at least 12 months at the date of inclusion in the study.
  * Subjects have to be registered in a general practitioner practice classified as 'up to standard' for at least 12 months at the date of inclusion in the study.
* Particular Case of New Born Children.

  * To ensure inclusion of subjects less than 1 year of age, they will be included regardless their observation time in CPRD.
* Inclusion Date

  * Inclusion criteria will be assessed for each calendar year between the Years 2000 and 2012.

Exclusion Criteria:

• For the analyses requiring the inclusion of HES data, HES records linked with more than one CPRD patient will be excluded from the analyses.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the subjects with diabetes mellitus diagnosed with hepatitis B, reported in the CPRD database of UK, from the Year 2000 to 2012.
Sampling Method: Non-Probability Sample
Enrollment: 161429 (Actual)
Dates: Start 2014-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of new HepB diagnosis among patients between 0-80 years of age previously diagnosed with DM, between 2000 and 2012, in the UK CPRD or Hospital Episodes Statistics (HES). | Up to 12 years
Occurrence of new HepB diagnosis among non-DM patients between 0-80 years of age, in the UK CPRD or HES. | Up to 12 years

SECONDARY OUTCOMES:
Hospitalisation episode recorded in HES due to HepB infection or complications among patients between 0-80 years of age previously diagnosed with DM and in DM-free (non-DM) patients, in the UK, for whom CPRD-HES linkage is available. | Up to 12 years
All cause mortality among HepB cases in the DM and DM-free (non-DM) patients between 0-80 years of age, in the UK. | Up to 12 years
HepB cause-specific mortality among DM and DM-free (non-DM) patients between 0-80 years of age, in the UK for whom CPRD-ONS mortality linkage is available. | Up to 12 years
New-onset or prevalent HepB diagnosis among new-onset or prevalent DM and DM-free (non-DM) patients between 0-80 years of age, in the UK, regardless of the onset of HepB in relation to the diagnosis of DM. | Up to 12 years

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Ferreira GLC, Marano C, De Moerlooze L, Guignard A, Feng Y, El Hahi Y, van Staa T. Incidence and prevalence of hepatitis B in patients with diabetes mellitus in the UK: A population-based cohort study using the UK Clinical Practice Research Datalink. J Viral Hepat. 2018 May;25(5):571-580. doi: 10.1111/jvh.12841. Epub 2018 Jan 17. PMID 29220868